CLINICAL TRIAL: NCT04558918
Title: A Randomized, Multicenter, Active-comparator Controlled, Open-label Trial to Evaluate Efficacy and Safety of Oral, Twice Daily LNP023 in Adult Patients With PNH and Residual Anemia, Despite Treatment With an Intravenous Anti-C5 Antibody.
Brief Title: Study of Efficacy and Safety of Twice Daily Oral LNP023 in Adult PNH Patients With Residual Anemia Despite Anti-C5 Antibody Treatment
Acronym: APPLY-PNH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023C12302; 2019-004665-40 (EudraCT Number)
Record Dates: First submitted 2020-08-27; First posted 2020-09-22 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: Paroxysmal nocturnal hemoglobinuria; Hemoglobin; Anemia; LNP023; eculizumab; ravulizumab
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Anemia | interventions — iptacopan; eculizumab; ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LNP023 200mg b.i.d. (Experimental): Iptacopan 200mg b.i.d. hard gelatin capsule. After 24 weeks of LNP023 200mg b.i.d. treatment in the Randomized Treatment Period, participants had the option to enter the Extension Treatment Period to receive an additional 24 weeks of LNP023 200mg b.i.d.
  Interventions: Drug: LNP023
- Anti-C5 antibody (Active Comparator): In the Randomized Treatment Period patients randomized to receive Anti-C5 antibody continued with the same stable regimen of Anti-C5 antibody therapy as they had received prior to randomization. For eculizumab (administered as intravenous infusion every 2 weeks), the maintenance dose was a fixed dose, whereas for ravulizumab (administered as intravenous infusion every 8 weeks), the maintenance dose was based on body weight. After 24 weeks of Anti-C5 antibody treatment in the Randomized Treatment Period, participants had the option to enter the Extension Treatment Period to receive 24 weeks of LNP023 200mg b.i.d.
  Interventions: Drug: Eculizumab; Drug: Ravulizumab

INTERVENTIONS:
Drug: LNP023 — Taken Orally b.i.d. Dosage Supplied: 200 mg Dosage form: Hard gelatin capsule Route of Administration: Oral
  Other Names: iptacopan
  Arms: LNP023 200mg b.i.d.
Drug: Eculizumab — Administered as intravenous infusion every 2 weeks as per the stable regimen, the maintenance dose is a fixed dose.
  Dosage Supplied: 300 mg/30mL Dosage form: Concentrate solution for infusion
  Arms: Anti-C5 antibody
Drug: Ravulizumab — Administered as intravenous infusion every 8 weeks, the maintenance dose is based on body weight.
  Dosage Supplied: 300 mg/30mL Dosage form: Concentrate solution for infusion
  Arms: Anti-C5 antibody

SUMMARY:
This study was a multi-center, randomized, open-label, active comparator-controlled, parallel group study.

The purpose of this Phase 3 study in PNH patients presenting with residual anemia despite treatment with anti-C5 antibody, was to determine whether iptacopan is efficacious and safe for the treatment of PNH through demonstration of superiority of iptacopan compared to anti-C5 antibody treatment.

DETAILED DESCRIPTION:
The study comprised three periods:

* A screening period lasting up to 8 weeks (unless there was a need to extend it for vaccinations required for inclusion, vaccinations were started as early as possible to avoid extension of the screening period)
* A 24-week randomized, open-label, active controlled, treatment period for the primary efficacy and safety analyses. Patients who met the eligibility criteria at screening were stratified based on the type of prior anti-C5 antibody treatment (eculizumab or ravulizumab) and based on the transfusion history as reported during the last 6 months prior to randomization (i.e. transfusion received/not received). Patients were randomized to one of the two treatment groups in an 8:5 ratio to either iptacopan monotherapy at a dose of 200 mg orally b.i.d. or i.v. anti-C5 antibody treatment (patients continued with the same regimen during the randomized treatment period as they were prior to randomization), respectively.
* A 24-week open-label, iptacopan treatment extension period. The patients randomized to the active comparator group were offered to switch to iptacopan on Day 168 (Week 24 visit) and entered the treatment extension period, after receiving a last dose of anti-C5 antibody treatment (eculizumab or ravulizumab). For patients in the comparator group not agreeing to switch treatment, Week 24 visit was the End of Study visit for the trial with no participation in the treatment extension period. For patients agreeing to switch to oral iptacopan, the Extension treatment started on the day after completion of the Week 24 visit. The patients in the iptacopan group who, in the opinion of investigator, benefitted from treatment and were taking iptacopan at Week 24 visit (i.e. did not permanently discontinue study medication), were offered the opportunity to continue oral iptacopan treatment during the treatment extension period.
* Data cut-off date used for the primary results submission was 26- Sep-2022

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ≥ 18 years of age with a diagnosis of PNH confirmed by high-sensitivity flow cytometry with clone size ≥ 10%
* Stable regimen of anti-C5 antibody treatment (either eculizumab or ravulizumab) for at least 6 months prior to randomization
* Mean hemoglobin level <10 g/dL
* Vaccination against Neisseria meningitidis infection is required prior to the start of treatment.
* If not received previously, vaccination against Streptococcus pneumoniae and Haemophilus influenzae infections should be given

Exclusion Criteria:

* Participants on a stable eculizumab dose but with a dosing interval of 11 days or less or patients on stable ravulizumab dose but with a dosing interval of less than 8 weeks.
* Known or suspected hereditary complement deficiency at screening
* History of hematopoietic stem cell transplantation
* Patients with laboratory evidence of bone marrow failure (reticulocytes <100x10E9/L; platelets <30x10E9/L; neutrophils <500x10E6/L).
* Active systemic bacterial, viral (incl. COVID-19), or fungal infection within 14 days prior to study drug administration
* A history of recurrent invasive infections caused by encapsulated organisms, e.g. meningococcus or pneumococcus.
* Major concurrent comorbidities including but not limited to severe kidney disease (e.g., eGFR < 30 mL/min/1.73 m2, dialysis), advanced cardiac disease (e.g., NYHA class IV), severe pulmonary disease (e.g., severe pulmonary hypertension (WHO class IV)), or hepatic disease (e.g., active hepatitis) that in the opinion of the investigator precludes participant's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (39):
- United States (5):
  - City Of Hope National Med Center City of Hope Medical Center, Duarte, California
  - Univ Cali Irvine ALS Neuromuscular, Orange, California
  - Augusta University Georgia Patient Treatment, Augusta, Georgia
  - Levine Cancer Insitute Carolinas Healthcare System, Charlotte, North Carolina
  - Cleveland Clinic Foundation Dept.ofTaussigCancer Center, Cleveland, Ohio
- Brazil (2):
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Ostrava, Poruba, Czechia
- France (3):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (5):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Riesa
  - Novartis Investigative Site, Ulm
- Italy (7):
  - Novartis Investigative Site, Ascoli Piceno, AP
  - Novartis Investigative Site, Avellino, AV
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Bassano del Grappa, VI
- Japan (7):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Suwa, Nagano
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Kyoto
- Novartis Investigative Site, Nijmegen, Netherlands
- Novartis Investigative Site, Seoul, South Korea
- Spain (3):
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
- Taiwan (2):
  - Novartis Investigative Site, Hualien City
  - Novartis Investigative Site, Taipei
- United Kingdom (2):
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] DeCastro C, Sheinberg P, Han B, Vallow S, Bermann G, Dhalke M, Kumar R, Dickie G, Galipeau N, Lamoureux R, Rupinski K, Lowe C, Nieves A, de Fontbrune FS, de Latour RP. Patient-Reported Meaningful Change in Symptoms and Impacts of Paroxysmal Nocturnal Hemoglobinuria (PNH) in Three Phase III Clinical Trials of Iptacopan. Patient. 2025 Nov;18(6):699-712. doi: 10.1007/s40271-025-00755-5. Epub 2025 Jul 22. PMID 40694294
- [Derived] Risitano AM, Kulasekararaj AG, Scheinberg P, Roth A, Han B, Maciejewski JP, Ueda Y, de Castro CM, Di Bona E, Fu R, Zhang L, Griffin M, Langemeijer SMC, Panse J, Schrezenmeier H, Barcellini W, Mauad VAQ, Schafhausen P, Tavitian S, Beggiato E, Chew LP, Gaya A, Huang WH, Jang JH, Kitawaki T, Kutlar A, Notaro R, Pullarkat V, Schubert J, Terriou L, Uchiyama M, Lee LWL, Yap ES, Frieri C, Marano L, de Fontbrune FS, Gandhi S, Trikha R, Alashkar F, Yang C, Liu H, Kelly RJ, Hochsmann B, Lawniczek T, Mahajan N, Solar-Yohay S, Kerloeguen C, Ferber P, Kumar R, Wang Z, Thorburn C, Maitra S, Li S, Verles A, Dahlke M, de Latour RP. Oral iptacopan monotherapy in paroxysmal nocturnal haemoglobinuria: final 48-week results from the open-label, randomised, phase 3 APPLY-PNH trial in anti-C5-treated patients and the open-label, single-arm, phase 3 APPOINT-PNH trial in patients previously untreated with complement inhibitors. Lancet Haematol. 2025 Jun;12(6):e414-e430. doi: 10.1016/S2352-3026(25)00081-X. PMID 40447351
- [Derived] Peffault de Latour R, Roth A, Kulasekararaj AG, Han B, Scheinberg P, Maciejewski JP, Ueda Y, de Castro CM, Di Bona E, Fu R, Zhang L, Griffin M, Langemeijer SMC, Panse J, Schrezenmeier H, Barcellini W, Mauad VAQ, Schafhausen P, Tavitian S, Beggiato E, Chew LP, Gaya A, Huang WH, Jang JH, Kitawaki T, Kutlar A, Notaro R, Pullarkat V, Schubert J, Terriou L, Uchiyama M, Wong Lee Lee L, Yap ES, Sicre de Fontbrune F, Marano L, Alashkar F, Gandhi S, Trikha R, Yang C, Liu H, Kelly RJ, Hochsmann B, Kerloeguen C, Banerjee P, Levitch R, Kumar R, Wang Z, Thorburn C, Maitra S, Li S, Verles A, Dahlke M, Risitano AM. Oral Iptacopan Monotherapy in Paroxysmal Nocturnal Hemoglobinuria. N Engl J Med. 2024 Mar 14;390(11):994-1008. doi: 10.1056/NEJMoa2308695. PMID 38477987
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2142

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 39 investigative sites in 12 countries: Netherlands(1), Germany(5), France(3), Japan(7), Korea, Republic of(1), Italy(7), Spain(3), Taiwan(2), United Kingdom(2), Czech Republic(1), United States(5), Brazil(2)
Pre-assignment Details: Vaccination against Neisseria meningitidis, Streptococcus pneumoniae and Haemophilus influenzae infections was required prior to the start of treatment, if the patient had not been previously vaccinated, or if a booster was required. The vaccines were given according to local regulations, at least 2 weeks prior to first dosing. If iptacopan treatment had to start earlier than 2 weeks post vaccination, prophylactic antibiotic treatment was initiated.
Period: Randomized Treatment Period
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Started | 62 | 35
Completed (completed the randomized treatment period) | 62 | 35
Not Completed | 0 | 0
Period: Extension Treatment Period
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Started | 61 | 34
Full Analysis Set (Includes all patients to whom study treatment has been assigned by randomization) | 62 | 35
Combined Full Analysis Set (Includes all patients randomized to LNP023 200 mg b.i.d and all patientsrandomized to anti-C5 treatment and who switched to LNP023 in the treatment extension period.) | 62 | 34
Completed (Completed the extension treatment period) | 61 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody | Total
Number analyzed (Participants) | 62 | 35 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (16.94) | 49.8 (16.69) | 51.0 (16.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 24 | 67
  Male | 19 | 11 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48 | 26 | 74
  Black or African American | 2 | 2 | 4
  Asian | 12 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Marginal Proportion (Expressed as Percentages) of Participants With Sustained Increase in Hemoglobin Levels From Baseline of ≥ 2 g/dL in the Absence of Red Blood Cell Transfusions
Description: Sustained increase in hemoglobin levels (responder) is defined as an increase from baseline in hemoglobin levels ≥ 2 g/dL on three out of four measurements taken at the visits occurring in last six weeks (between Day 126 and 168) of the randomized treatment period, without requiring red blood cell (RBC) transfusions between Day 14 and Day 168. Requiring RBC transfusions refers to any patient receiving transfusions or meeting protocol defined criteria (Hemoglobin level ≤ 9 g/dL with signs /and or symptoms of sufficient severity to warrant a transfusion or Hemoglobin of ≤ 7 g/dL, regardless of presence of clinical signs and/or symptoms).
  The term 'marginal proportion' can be interpreted as the population average probability of being a responder for each treatment group. These values include adjustment for baseline covariates and missing data has also been taken into account.
Time Frame: Baseline, hemoglobin between Day 126 and Day 168 and absence of transfusions between Day 14 and Day 168
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 62 | 35
Percentage of responders | 82.3 [73.4 to 90.2] | 2.0 [1.1 to 4.0]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Superiority; p < 0.0001, Regression, Logistic — two sided unadjusted p-value; Logistic regression model using Firth; Odds Ratio (OR) = 338.25, 95% CI 2-sided [25.07 to 4564.14]
Statistical Analysis 2: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Superiority; Difference in marginal proportion = 80.2, 95% CI 2-sided [71.2 to 87.6]

2. Primary Outcome: Marginal Proportion (Expressed as Percentages) of Participants With Sustained Hemoglobin Levels of ≥ 12 g/dL in the Absence of Red Blood Cell Transfusions
Description: Sustained hemoglobin levels (responder) is defined as hemoglobin levels ≥ 12 g/dL on three out of four measurements taken at the visits occurring in last six weeks (between Day 126 and 168) of the randomized treatment period, without requiring red blood cell (RBC) transfusions between Day 14 and Day 168. Requiring RBC transfusions refers to any patient receiving transfusions or meeting protocol defined criteria (Hemoglobin level ≤ 9 g/dL with signs /and or symptoms of sufficient severity to warrant a transfusion or Hemoglobin of ≤ 7 g/dL, regardless of presence of clinical signs and/or symptoms).
  The term 'marginal proportion' can be interpreted as the population average probability of being a responder for each treatment group. These values include adjustment for baseline covariates and missing data has also been taken into account.
Time Frame: Hemoglobin between Day 126 and Day 168 and absence of transfusions between Day 14 and Day 168
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 62 | 35
Percentage of responders | 68.8 [58.4 to 78.9] | 1.8 [0.9 to 4.0]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Superiority; p < 0.0001, Regression, Logistic — two sided unadjusted p-value; Logistic regression model using Firth; Odds Ratio (OR) = 495.74, 95% CI 2-sided [24.41 to 10066.53]
Statistical Analysis 2: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Superiority; Diff. in marginal proportion = 67.0, 95% CI 2-sided [56.4 to 76.9]

3. Primary Outcome: Percentage of Patients Meeting Hematological Response Criterion After the Start of LNP023 Treatment
Description: Patients with hematological response are those with ≥ 2g/dL increase in hemoglobin from baseline regardless of transfusions and patients with Hb ≥ 12g/dL regardless of transfusions.
  Patients in the LNP023-LNP023 group received iptacopan from Day 1 to Day 336 (48 weeks) while patients in the anti-C5 antibody-LNP023 group received iptacopan from Day 169 to Day 336 (treatment extension period - 24 weeks).
Time Frame: Up to 48 weeks
Population: Combined Full Analysis Set: includes all patients randomized to LNP023 200 mg b.i.d and all patients randomized to anti-C5 treatment and who switched to LNP023 in the treatment extension period.
Measure: Number; unit: Percentage of participants
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 62 | 34
Percentage of participants
  ≥2 g/dL increase in Hb from baseline irrespective of RBC transfusions | 86.4 | 72.4
  Hb ≥12 g/dL irrespective of RBC transfusions | 67.8 | 58.6

4. Primary Outcome: Number of Patients Not Requiring RBC Transfusions After the Start of LNP023 Treatment
Description: Requiring RBC transfusions refers to any patient receiving transfusions or meeting protocol defined criteria (Hemoglobin level ≤ 9 g/dL with signs /and or symptoms of sufficient severity to warrant a transfusion or Hemoglobin of ≤ 7 g/dL, regardless of presence of clinical signs and/or symptoms).
  Patients randomized to anti-C5 treatment switched to LNP023 (iptacopan) on Day 169 and were treated until Day 336 (treatment extension period).
Time Frame: Up to 48 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 62 | 34
Participants
  Since Day 1 of LNP023 treatment | 51 | 31
  Since Day 14 of LNP023 treatment | 57 | 32

5. Primary Outcome: Change From Baseline in Hemoglobin at Visit Day 336
Description: Patients randomized to anti-C5 treatment switched to LNP023 (iptacopan) on Day 169 and were treated until Day 336 (treatment extension period).
Time Frame: Baseline, Day 336
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization. Only participants with valid HB measurements at baseline and Day 336 were analyzed.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 59 | 30
g/dL | 3.35 [3.04 to 3.67] | 3.36 [2.94 to 3.79]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Other; Adjusted mean difference = -0.01, 95% CI 2-sided [-0.53 to 0.51]

6. Primary Outcome: Change From Baseline in FACIT-Fatigue Questionnaire at Day 336
Description: The FACIT-Fatigue is a 13-item questionnaire with support for its validity and reliability in PNH that assesses patient self-reported fatigue and its impact on daily activities and function. All FACIT scales are scored so that a high score is better. As each of the 13 items of the FACIT-F Scale ranges from 0-4, the range of possible scores is 0-52, with 0 being the worst possible score and 52 the best.
  Patients randomized to anti-C5 treatment switched to LNP023 (iptacopan) on Day 169 and were treated until Day 336 (treatment extension period).
Time Frame: Baseline, Day 336
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization. Only participants with valid FACIT-Fatigue scores at baseline and Day 336 were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 55 | 26
score on a scale | 9.80 [8.04 to 11.56] | 10.96 [8.58 to 13.34]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Other; Adjusted mean difference = -1.17, 95% CI 2-sided [-4.01 to 1.68]

7. Secondary Outcome: Marginal Proportion (Expressed as Percentages) of Participants Who Remain Free From Transfusions
Description: Marginal proportion (expressed as percentages) of participants who did not require transfusions between Day 14 and Day 168. Requiring red blood cell transfusions refers to any patient receiving transfusions or meeting protocol defined criteria (Hemoglobin level ≤ 9 g/dL with signs /and or symptoms of sufficient severity to warrant a transfusion or Hemoglobin of ≤ 7 g/dL, regardless of presence of clinical signs and/or symptoms). The term 'marginal proportion' can be interpreted as the population average probability of being a responder for each treatment group. These values include adjustment for baseline covariates and missing data has also been taken into account.
Time Frame: Between Day 14 and Day 168
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 62 | 35
Percentage of participants | 94.8 [88.1 to 100.0] | 25.9 [11.6 to 42.4]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Superiority; p < 0.0001, Conditional logistic regression — two sided unadjusted p-value; Odds Ratio (OR) = 108.41, 95% CI 2-sided [17.25 to 681.24]
Statistical Analysis 2: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; logistic regression model; Test type: Superiority; Diff. in marginal proportion = 68.9, 95% CI 2-sided [51.4 to 83.9]

8. Secondary Outcome: Change From Baseline in Hemoglobin Between Day 126 and 168
Description: Change from baseline in hemoglobin levels as mean of visits between Day 126 and Day 168.
  For this analysis, in order to factor out the effect of transfusions, if a patient had a transfusion during the randomized treatment period, then the hemoglobin values 30 days following the transfusion were excluded and hemoglobin data were imputed.
Time Frame: Baseline and mean of visits between Day 126 and 168
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 62 | 35
g/dL | 3.60 [3.33 to 3.88] | -0.06 [-0.45 to 0.34]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Superiority; p < 0.0001, Mixed Model of Repeated Measures (MMRM) — two sided unadjusted p-value; Adjusted mean diff. = 3.66, 95% CI 2-sided [3.20 to 4.12]

9. Secondary Outcome: Change From Baseline in FACIT-Fatigue Questionnaire in the Randomized Treatment Period
Description: The FACIT-Fatigue is a 13-item questionnaire with support for its validity and reliability in PNH that assesses patient self-reported fatigue and its impact on daily activities and function. All FACIT scales are scored so that a high score is better. As each of the 13 items of the FACIT-F Scale ranges from 0-4, the range of possible scores is 0-52, with 0 being the worst possible score and 52 the best.
Time Frame: Baseline, mean of visits between Day 126 and Day 168
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization. Only participants with valid FACIT-Fatigue scores at baseline and between day 126 and day 168 were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 62 | 33
score on a scale | 8.59 [6.72 to 10.47] | 0.31 [-2.20 to 2.81]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Superiority; p < 0.0001, Mixed Model of Repeated Measures (MMRM) — two sided unadjusted p-value; Mean Difference (Net) = 8.29, 95% CI 2-sided [5.28 to 11.29]

10. Secondary Outcome: Change From Baseline in Absolute Reticulocyte Count in the Randomized Treatment Period
Description: Change from baseline in absolute reticulocyte count as mean of visits between Day 126 and Day 168
Time Frame: Baseline and mean of visits between Day 126 and 168
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization.
Measure: Mean (95% Confidence Interval); unit: x10^9 cells/L
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 62 | 35
x10^9 cells/L | -115.81 [-126.40 to -105.23] | 0.34 [-13.04 to 13.72]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Superiority; p < 0.0001, Mixed Model of Repeated Measures (MMRM) — two sided unadjusted p-value; Mean Difference (Net) = -116.15, 95% CI 2-sided [-132.04 to -100.26]

11. Secondary Outcome: Ratio to Baseline in Log-transformed LDH in the Randomized Treatment Period
Description: Average of the Lactate dehydrogenase (LDH) log transformed ratio to baseline in each treatment estimated between Day 126 and Day 168.The log transformation used refers to the natural log (base of e).
Time Frame: Baseline and mean of visits between Day 126 and 168
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization.
Measure: Geometric Mean (95% Confidence Interval); unit: ln(ratio)
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 62 | 35
ln(ratio) | 0.96 [0.90 to 1.03] | 0.98 [0.89 to 1.07]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Superiority; p = 0.8361, Mixed Model of Repeated Measures (MMRM) — two sided unadjusted p-value; Geometric mean ratio = 0.99, 95% CI 2-sided [0.89 to 1.10]

12. Secondary Outcome: Adjusted Annualized Clinical BTH Rate in the Randomized Treatment Period
Description: Adjusted annualized rate of clinical breakthrough hemolysis (BTH) events are from negative binomial model.
  A patient with multiple occurrences of an event under one treatment is counted only once for that treatment.
  The breakthrough is defined clinical if either there is a decrease in hemoglobin levels equal to or more than 2 g/dL (compared to the latest assessment, or within 15 days) or if patients present signs or symptoms of gross hemoglobinuria, painful crisis, dysphagia or any other significant clinical PNH-related signs & symptoms, in presence of laboratory evidence of intravascular hemolysis.
Time Frame: Between Day 1 and Day 168
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: BTH events/year
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 62 | 35
BTH events/year | 0.07 [0.02 to 0.31] | 0.67 [0.26 to 1.72]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Superiority; p = 0.01183, Negative binomial model — two sided unadjusted p-value; Rate ratio = 0.10, 95% CI 2-sided [0.02 to 0.61]
Statistical Analysis 2: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Superiority; Rate difference = -0.60, 95% CI 2-sided [-1.24 to 0.04]

13. Secondary Outcome: Adjusted Annualized Major Adverse Vascular Events Rate in the Randomized Treatment Period
Description: Adjusted annualized Major Adverse Vascular Events (MAVEs incl. thrombosis) rate. A MAVE is defined as: acute peripheral vascular occlusion, amputation (non-traumatic; nondiabetic), cerebral arterial occlusion/cerebrovascular accident, cerebral venous occlusion, dermal thrombosis, gangrene (non-traumatic; nondiabetic), hepatic/portal vein thrombosis (Budd-Chiari syndrome), mesenteric/visceral arterial, thrombosis or infarction, mesenteric/visceral vein thrombosis or infarction, myocardial infarction, pulmonary embolus, renal arterial thrombosis, renal vein thrombosis, thrombophlebitis / deep vein thrombosis, transient ischemic attack, unstable angina or other.
  A patient with multiple occurrences of an event under one treatment is counted only once for that treatment.
Time Frame: Between Day 1 and Day 168
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization.
Measure: Number (95% Confidence Interval); unit: MAVE events/year
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 62 | 35
MAVE events/year | 0.03 [0.00 to 0.25] | 0.00 [0.00 to 0.00]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Superiority; p = 0.31731, Poisson model — two sided unadjusted p-value; rate difference = 0.03, 95% CI 2-sided [-0.03 to 0.10]

14. Other Pre Specified Outcome: Change From Baseline in Absolute Reticulocyte Count at Day 336
Description: Change from baseline in absolute reticulocyte count at visit Day 336. Patients randomized to anti-C5 antibody were switched to LNP023 (iptacopan) on Day 169 and were treated until Day 336 (treatment extension period).
Time Frame: Baseline and Day 336
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization. Only participants with valid absolute reticulocyte count at baseline and Day 336 were analyzed.
Measure: Mean (95% Confidence Interval); unit: x10^9 cells/L
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 57 | 30
x10^9 cells/L | -106.26 [-117.57 to -94.96] | -107.95 [-123.18 to -92.73]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Other; Adjusted mean difference = 1.69, 95% CI 2-sided [-16.86 to 20.23]

15. Other Pre Specified Outcome: Ratio to Baseline in Log-transformed LDH at Visit Day 336
Description: Average of the Lactate dehydrogenase (LDH) log transformed ratio to baseline at visit Day 336.The log transformation used refers to the natural log (base of e).
  Patients randomized to anti-C5 treatment switched to LNP023 (iptacopan) on Day 169 and were treated until Day 336 (treatment extension period).
Time Frame: Baseline and Day 336
Population: Full Analysis Set (FAS): patients to whom study treatment had been assigned by randomization. Only participants with valid LDH measurements at baseline and Day 336 were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ln(ratio)
Arm/Group | LNP023 200mg b.i.d. | Anti-C5 Antibody
Number analyzed (Participants) | 61 | 33
ln(ratio) | 1.11 [1.02 to 1.22] | 0.99 [0.88 to 1.11]
Statistical Analysis 1: Comparison: LNP023 200mg b.i.d. vs Anti-C5 Antibody; Test type: Other; Geometric mean ratio = 1.12, 95% CI 2-sided [0.97 to 1.30]

16. Primary Outcome: Adjusted Annualized Clinical BTH Rate After the Start of LNP023 Treatment
Description: This endpoint is considering clinical BTH events after the start of LNP023 treatment. Therefore, results are presented in a single arm on LNP023 since it includes all patients in the Combined Full analysis set.
  Adjusted annualized rate of clinical breakthrough hemolysis (BTH) events are from negative binomial model. A patient with multiple occurrences of an event under one treatment is counted only once for that treatment.The breakthrough is defined clinical if either there is a decrease in hemoglobin levels equal to or more than 2 g/dL (compared to the latest assessment, or within 15 days) or if patients present signs or symptoms of gross hemoglobinuria, painful crisis, dysphagia or any other significant clinical PNH-related signs & symptoms, in presence of laboratory evidence of intravascular hemolysis.
Time Frame: Up to 336 Days
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: BTH events/year
Groups:
- Overall LNP023 200 mg b.i.d During the Entire Study: Includes all patients randomized to LNP023 200 mg b.i.d and all patients randomized to anti-C5 treatment and who switched to LNP023 in the treatment extension period
Arm/Group | Overall LNP023 200 mg b.i.d During the Entire Study
Number analyzed (Participants) | 96
BTH events/year | 0.11 [0.05 to 0.23]

17. Primary Outcome: Adjusted Annualized Major Adverse Vascular Events Rate After the Start of LNP023 Treatment
Description: This endpoint is considering clinical BTH events after the start of LNP023 treatment. Therefore, results are presented in a single arm on LNP023 since it includes all patients in the Combined Full analysis set.
  Adjusted annualized Major Adverse Vascular Events (MAVEs incl. thrombosis) rate. A MAVE is defined as: acute peripheral vascular occlusion, amputation (non-traumatic; nondiabetic), cerebral arterial occlusion/cerebrovascular accident, cerebral venous occlusion, dermal thrombosis, gangrene (non-traumatic; nondiabetic), hepatic/portal vein thrombosis (Budd-Chiari syndrome), mesenteric/visceral arterial, thrombosis or infarction, mesenteric/visceral vein thrombosis or infarction, myocardial infarction, pulmonary embolus, renal arterial thrombosis, renal vein thrombosis, thrombophlebitis / deep vein thrombosis, transient ischemic attack, unstable angina or other.
  A patient with multiple occurrences of an event under one treatment is counted only once for that treatment.
Time Frame: Up to 336 Days
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: MAVE events/year
Arm/Group | Overall LNP023 200 mg b.i.d During the Entire Study
Number analyzed (Participants) | 96
MAVE events/year | 0.04 [0.01 to 0.13]

ADVERSE EVENTS:
Time Frame: Adverse events of LNP023 group were reported from first dose of study treatment until the end of study treatment plus 30 days, up to a maximum duration of 48 weeks
Description: Adverse events of anti-C5 antibody were reported from the date of first administration of anti-C5 study treatment in the randomized treatment period to the date of the last actual administration of anti-C5 antibody in the randomized treatment period.
Groups:
- LNP023 200mg b.i.d. (Randomized Treatment Period): Patients who were randomized to LNP023 200mg b.i.d. (time frame is up to week 24)
- Anti-C5 Antibody (Randomized Treatment Period): Patients who were randomized to Anti-C5 antibody (time frame is up to week 24)
- LNP023 200mg b.i.d. (Randomized Treatment Period + Extension Treatment Period): Patients who were randomized LNP023 200mg b.i.d. (time frame is up to week 48)
- Any LNP023 200mg b.i.d. (Randomized Treatment Period + Extension Treatment Period): Patients who were randomized to LNP023 200mg b.i.d. and patients who switched from Anti-C5 antibody to LNP023 200mg b.i.d. (time frame is up to 48 weeks)
Arm/Group | LNP023 200mg b.i.d. (Randomized Treatment Period) | Anti-C5 Antibody (Randomized Treatment Period) | LNP023 200mg b.i.d. (Randomized Treatment Period + Extension Treatment Period) | Any LNP023 200mg b.i.d. (Randomized Treatment Period + Extension Treatment Period)
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/35 | 0/62 | 0/96
Serious Adverse Events (participants affected / at risk) | 6/62 | 5/35 | 9/62 | 13/96
Other Adverse Events (participants affected / at risk) | 34/62 | 21/35 | 43/62 | 62/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNP023 200mg b.i.d. (Randomized Treatment Period) (N=62) | Anti-C5 Antibody (Randomized Treatment Period) (N=35) | LNP023 200mg b.i.d. (Randomized Treatment Period + Extension Treatment Period) (N=62) | Any LNP023 200mg b.i.d. (Randomized Treatment Period + Extension Treatment Period) (N=96)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Extravascular haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 1 | 1
Pancreatolithiasis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 2 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 1
Systemic infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0 | 1 | 1
Influenza A virus test positive (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Bilirubinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LNP023 200mg b.i.d. (Randomized Treatment Period) (N=62) | Anti-C5 Antibody (Randomized Treatment Period) (N=35) | LNP023 200mg b.i.d. (Randomized Treatment Period + Extension Treatment Period) (N=62) | Any LNP023 200mg b.i.d. (Randomized Treatment Period + Extension Treatment Period) (N=96)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 2 | 6 | 6 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 9 | 2 | 10 | 12
Nausea (Gastrointestinal disorders) | 6 | 1 | 8 | 11
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2 | 5
Pyrexia (General disorders) | 2 | 3 | 4 | 5
COVID-19 (Infections and infestations) | 4 | 7 | 17 | 25
Nasopharyngitis (Infections and infestations) | 7 | 3 | 9 | 12
Sinusitis (Infections and infestations) | 2 | 3 | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 3 | 4
Urinary tract infection (Infections and infestations) | 4 | 1 | 7 | 7
Blood lactate dehydrogenase increased (Investigations) | 4 | 3 | 6 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 7 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 3
Dizziness (Nervous system disorders) | 4 | 0 | 4 | 4
Headache (Nervous system disorders) | 11 | 1 | 12 | 14
Insomnia (Psychiatric disorders) | 3 | 0 | 4 | 4
Hypertension (Vascular disorders) | 3 | 0 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT04558918/Prot_003.pdf
  • Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT04558918/SAP_001.pdf